CLINICAL TRIAL: NCT05612490
Title: Evaluation of the Furosemide Stress Test to Predict Successful Liberation From Renal Replacement Therapy in Critically Ill Patients
Brief Title: Furosemide Stress Test to Predict Successful Liberation From RRT
Acronym: FST-RRT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antoine Schneider, Doctor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2022-01826
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury
Keywords: Renal replacement therapy; Acute Kidney Injury; Furosemide Stress Test
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sample at D0, D1, D2 and D3 and on RRT restart (if applicable)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically ill patients undergoing RRT: Patients admitted to participating ICU and receiving renal replacement therapy.
  Interventions: Drug: Furosemide stress test

INTERVENTIONS:
Drug: Furosemide stress test — The FST corresponds to the intravenous single-dose administration of 1 mg/kg (1.5 mg/kg in previously exposed patients) of furosemide and the assessment of resulting diuresis in the following two hours. In the 12 hours following the first RRT liberation, a FST will be performed. The test will be considered positive if urinary output is ≥200 mL in the two hours following furosemide administration.
  Other Names: FST

SUMMARY:
The proposed study will evaluate if a standardised dose of furosemide administered in the 12 hours after RRT liberation can predict successful liberation in critically ill patients. The dose that will be administered is in accordance with the prescribing information.

DETAILED DESCRIPTION:
Response to furosemide administration is commonly used in clinical practice to assess a patient's potential for RRT liberation. However, this administration is not standardized and practices varies greatly. Rapid recognition of unsuccessful RRT liberation is crucial to avoid further complications such as fluid overload or acid-base and electrolyte disorders. The FST corresponds to the intravenous administration of 1 mg/kg (1.5 mg/kg in previously exposed patients) of furosemide and the assessment of resulting diuresis in the following two hours. FST is able to predict progression from AKI stage I and II to stage III with a high sensitivity (87.1%) and specificity (84.1%), area under the ROC curve 0.87. However, the ability of FST to predict RRT liberation has never been formally assessed.

ELIGIBILITY:
Inclusion Criteria:

* Receiving continuous or intermittent RRT for AKI
* Having an indwelling urinary catheter
* Clinical decision by physician in charge to attempt RRT liberation
* lnformed consent signed by the patient himself / legal representative or authorization received from independent physician

Exclusion Criteria:

* Electrolyte disturbances or hemodynamic instability precluding the use of furosemide (sodium > 155 mmol/L and/or potassium < 3.0 mmol/L and/or metabolic alkalosis > 7.50 and/or mean arterial pressure < 60 mmHg)
* Known furosemide allergy
* Urine output ≥ 100 mL/h for at least two hours
* Recent (< 24 hours) FST
* Known end-stage chronic renal disease at ICU admission
* Withdrawal of life support decision taken before inclusion
* Patient already participating in conflicting research study
* Patient having already participated in this current study
* Any other contraindication of furosemide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients receiving continuous RRT for AKI
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Successful liberation of RRT within 72 hours after FST | within 72 hours
  No renal replacement therapy administered

SECONDARY OUTCOMES:
Successful liberation of RRT at ICU discharge | At time of ICU discharge, assessed up to 90 days post inclusion
  No renal replacement therapy administered
Successful liberation of RRT at hospital discharge | At time of hospital discharge, assessed up to 90 days post inclusion
  No renal replacement therapy administered
Adverse events associated with the intervention | within 6 hours
  (electrolyte disturbances, hypotension)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Schneider, MD PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chawla LS, Davison DL, Brasha-Mitchell E, Koyner JL, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Kimmel PL, Seneff MG. Development and standardization of a furosemide stress test to predict the severity of acute kidney injury. Crit Care. 2013 Sep 20;17(5):R207. doi: 10.1186/cc13015. PMID 24053972